CLINICAL TRIAL: NCT02786615
Title: Increasing Involvement of MSM in the Continuum of Care in Kazakhstan
Brief Title: Increasing MSM in the Continuum of Care in Kazakhstan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elwin Wu, Associate Professor of Social Work, Columbia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAQ7251; 1R01DA040513-01A1 (NIH)
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: HIV; Substance-Related Disorders
Keywords: men who have sex with men (MSM)
MeSH Terms: conditions — Substance-Related Disorders; Homosexuality

STUDY DESIGN:
Intervention Model Description: Stepped-wedge design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer Unity (Experimental): Subjects assigned to this arm would receive a 4-session, group-delivered intervention focusing on peer/social network-based recruitment and referral program to receive HIV prevention and treatment services in the community.
  Interventions: Behavioral: Peer Unity
- Pre-implementation (No Intervention): Subjects assigned to this arm would not receive the group-delivered intervention.

INTERVENTIONS:
Behavioral: Peer Unity — A 4-session, group-delivered intervention focusing on peer/social network-based recruitment and referral program to receive HIV prevention and treatment services in the community.
  Arms: Peer Unity

SUMMARY:
This study addresses the disproportionate representation of men who have sex with men (MSM) in the human immunodeficiency virus/acquired immune deficiency syndrome (HIV/AIDS) pandemic in Kazakhstan, a country that has seen some of the largest growth in new HIV infections since the turn of the century. Using a stepped wedge trial across 3 cities in Kazakhstan, the proposed study will test a strategic and innovative social network-based intervention for MSM who use drugs in Kazakhstan as a strategy to increase their numbers in the HIV continuum of care.

DETAILED DESCRIPTION:
The intervention is designed to utilize MSM as experts and leverage social network processes to increase the number of MSM in Kazakhstan to be engaged in the HIV continuum of care. The unit of randomization will be a city, with the timing of roll-out of the social network-based intervention in each of the study's cities-Almaty, Nur-Sultan (formerly Astana), and Shymkent-under experimental control. Receipt/delivery of an intervention to enrolled participants will depend on whether the city is in the intervention delivery phase or not. If a participant is in a city during a time period where the intervention is not being delivered then for that time period, the participant is in the control condition. If the participant is in a city during a time period where the intervention is being delivered then the participant (in fact, all participants in that city) will be considered assigned to the intervention group at that time. In theory, all participants will have the opportunity to experience and receive the intervention. Some participants will be enrolled after the intervention has been rolled out in the city in which they reside; thus, they will only experience the intervention condition and not the control condition.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years old;
* identify as male; and
* report oral or anal intercourse with another man in the past 12 months; and
* report binge alcohol consumption and/or illicit use of substances in the past 12 months

Exclusion Criteria:

* has a language or cognitive impairment that would prevent comprehension of study procedures, risks, and benefits (described in Russian during the informed consent process)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 987 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Engagement in the HIV care continuum: HIV testing | Past 6 months
  Has participant received an HIV test in the past 6 months

SECONDARY OUTCOMES:
For PLWH, engagement in the HIV care continuum related to HIV medical treatment | Since confirmed HIV infection diagnosis
  For PLWH, visiting AIDS center, receiving ART, and/or achieving viral suppression (descriptive/exploratory due to limited statistical power given only a smaller fraction of sample will have known HIV infection)

CONTACTS AND LOCATIONS:
Overall Officials: Elwin Wu, PhD, Principal Investigator — Columbia University
Locations (2):
- Columbia University School of Social Work, New York, New York, United States
- Global Health Research Center of Central Asia, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared: (1) in accordance with journal requirements, and/or (2) via publicly accessible data repository (e.g., Academic Commons)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: With or after publication, in perpetuity

REFERENCES:
- [Derived] Reeder KG, Lee YG, Sung J, Vinogradov V, Zhakupova G, Mergenova G, Davis A, Paine EA, Primbetova S, Terlikbayeva A, Kali S, Hunt T, Wu E. Trans Health is Public Health: The Prevalence of HIV Among Trans and Gender Expansive People in Kazakhstan. Res Sq [Preprint]. 2024 Sep 24:rs.3.rs-5124958. doi: 10.21203/rs.3.rs-5124958/v1. PMID 39399678
- [Derived] Wu E, Lee YG, Vinogradov V, Zhakupova G, Mergenova G, Davis A, Paine EA, Hunt T, Reeder K, Primbetova S, Terlikbayeva A, Laughney C, Chang M, Baiserkin B, Abishev A, Tukeyev M, Abdraimov S, Denebayeva A, Kasymbekova S, Tazhibayeva G, Kozhakhmet M. Increasing HIV Testing Among Sexual and Gender Expansive Men in Kazakhstan: A Stepped-Wedge Randomized Trial of a Community-Level Intervention. medRxiv [Preprint]. 2024 Aug 2:2024.08.01.24311235. doi: 10.1101/2024.08.01.24311235. PMID 39132483